CLINICAL TRIAL: NCT00701142
Title: Haemocomplettan® P in Patients Experiencing Acute Bleeding While Undergoing Aortic Replacement Surgery
Brief Title: Haemocomplettan® P During Aortic Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1470; BI3023_2002 (Other: CSL Behring); 2007-004612-31 (EudraCT Number)
Record Dates: First submitted 2008-06-16; First posted 2008-06-19 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2011-02

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm | interventions — Fibrinogen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Haemocomplettan® P (Active Comparator): Intravenous infusion during aortic surgery
  Interventions: Biological: Haemocomplettan® P
- Saline solution (Placebo Comparator)
  Interventions: Biological: Saline solution

INTERVENTIONS:
Biological: Haemocomplettan® P — Single intravenous infusion
  Other Names: RiaSTAP
  Arms: Haemocomplettan® P
Biological: Saline solution — Single intravenous infusion
  Arms: Saline solution

SUMMARY:
The primary purpose is to show that administration of Haemocomplettan® P significantly reduces the amount of blood products needed during aortic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older
* Undergoing elective thoracoabdominal aortic replacement surgery (TAAA) or thoracic aortic replacement surgery (TAA)
* Understood and willingly given written informed consent (German language) to participate following an explanation of study background, restrictions, and procedures
* Experience clinically relevant bleeding of the microvasculature following removal of CPB during surgery

Exclusion Criteria:

* Positive pregnancy test, pregnancy or lactation
* Women of child bearing age not using a medically approved method of contraception during the study
* Previous aortic replacement at the same aortic site (redo surgeries)
* Undergoing an emergency operation
* Proof or suspicion of a congenital or acquired coagulation disorder (e.g. VWD or via severe liver disease)
* Myocardial Infarction (MI) or apoplexy in the 2 months preceding study surgery
* ASA administration in the 3 days preceding study surgery, and a pathological (<74.5 U) ASPI Multiplate® test immediately preceding surgery begin
* Clopidogrel administration in the 5 days preceding study surgery, and a pathological (<31.1 U) ADP/PG Multiplate® test immediately preceding surgery begin
* Tirofiban administration in the 2 days preceding study surgery, and a pathological (<94.1 U) TRAP Multiplate® test immediately preceding surgery begin
* Phenprocoumon administration in the 5 days preceding study surgery, and an INR > 1.28 immediately preceding surgery begin
* Participation in another clinical study in the 4 weeks preceding aortic replacement
* Sensitivity to any of the components of study medication, or to MPs with a similar chemical structure to any of the components of study medication
* Any indication that the restrictions or procedures of the study may not be adhered to (e.g. an uncooperative attitude)
* Any indication that the study restrictions, procedures, or consequences therein have not been considered or understood, such that informed consent cannot be convincingly given
* Multiple morbidities, with a notably constrained remaining length of life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Combined number of units of allogeneic blood products (platelets + FFP + RBCs) administered to subjects. | From administration of Haemocomplettan® P until 24 hours later

SECONDARY OUTCOMES:
Proportion of subjects that receive no allogeneic blood products (neither platelets, FFP, nor RBCs) | From administration of Haemocomplettan® P until 24 hours later
Duration of stay in ICU | Last suture of initial surgery to end of ICU stay
Duration of hospital stay | Last suture of initial surgery to end of hospital stay
Mortality | 45 days post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Niels Rahe-Meyer, Dr. Dr., Principal Investigator — Abteilung Anästhesiologie, Carl-Neuberg-Strasse 1 / K5, 30177 Hannover
Locations (1):
- Medical School Hannover (MHH), Hanover, Germany

REFERENCES:
- [Result] Rahe-Meyer N, Solomon C, Hanke A, Schmidt DS, Knoerzer D, Hochleitner G, Sorensen B, Hagl C, Pichlmaier M. Effects of fibrinogen concentrate as first-line therapy during major aortic replacement surgery: a randomized, placebo-controlled trial. Anesthesiology. 2013 Jan;118(1):40-50. doi: 10.1097/ALN.0b013e3182715d4d. Erratum In: Anesthesiology. 2013 May;118(5):1244. PMID 23249928
- [Derived] Rahe-Meyer N, Hanke A, Schmidt DS, Hagl C, Pichlmaier M. Fibrinogen concentrate reduces intraoperative bleeding when used as first-line hemostatic therapy during major aortic replacement surgery: results from a randomized, placebo-controlled trial. J Thorac Cardiovasc Surg. 2013 Mar;145(3 Suppl):S178-85. doi: 10.1016/j.jtcvs.2012.12.083. PMID 23410777
- [Derived] Schochl H, Posch A, Hanke A, Voelckel W, Solomon C. High-dose fibrinogen concentrate for haemostatic therapy of a major trauma patient with recent clopidogrel and aspirin intake. Scand J Clin Lab Invest. 2010 Oct;70(6):453-7. doi: 10.3109/00365513.2010.500396. PMID 20624109